CLINICAL TRIAL: NCT04761666
Title: Influence of Verticalization on Bone Mineral Density and Biological Parameters of Bone Remodeling in Children With Severe Cerebral Palsy
Acronym: CPABONE
Status: Withdrawn | Type: Observational
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0036
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Cerebral Palsy; Osteoporosis; Bone Mineral Density; Bone Remodeling Disorder; Fracture
Keywords: Cerebral Palsy; Osteoporosis; bone mineral density; bone remodelling factors; Fracture; static verticalization device; weight bearing exersices
MeSH Terms: conditions — Cerebral Palsy; Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- static verticalization device: children with severe cerebral palsy (GMFCS IV & V) with static verticalization device
- non verticalization device: children with severe cerebral palsy (GMFCS IV & V) without static verticalization device

SUMMARY:
Low bone mineral density affects 77% of children with severe cerebral palsy (GMFCS IV & V) with an increased fracture risk of 4%. One strategy supposed to improve bone mineral density is verticalisation with static devices. Nowadays there is no time recommendation of verticalisation however high intensity verticalisation has been shown to be effective in improving bone mineral density in childrens with cerebral palsy, but difficult to apply in real life due to lack of qualified therapists, device's complexity, and severe impairment in those children. The investigators aim to compare bone mineral density and bone remodelling factors of verticalized and non verticalized childrens with severe cerebral palsy as achieved in everyday life. The investigators conduced a retrospective study comparing bone mineral density and factors who influence bone remolling in severe cerebral palsy's according to whether they are verticalized or not.

ELIGIBILITY:
Inclusion Criteria:

* patients with cerebral palsy GMFCS (gross motor functional classification scale) IV-V
* age of patients 3-18 years

Exclusion Criteria:

* patients with neuro muscular disease
* patient age < 3 years old and > 18 years old
* patient with constitutionnal bone disease
* patient with growth hormone treatment
* patient with surgery < 6 months
* patient with fracture <3 months
* Refusal of the legal representative

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children whom age is between 3 and 18 years old. Children with cerebral palsy GMFCS (gross motor functionnal classification scale) IV-V.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Variation of Densitometric Z score between both groups | 6 months
  A Z-score compares the patient bone density to the average bone density of people your own age and gender.A Z-score is helpful in diagnosing secondary osteoporosis and is always used for children. It is most useful when the score is less than 2 standard deviations below this normal. In this setting, it is helpful to scrutinize for coexisting illnesses or treatments that may contribute to osteoporosis such as glucocorticoid therapy, hyperparathyroidism, or alcoholism.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No